CLINICAL TRIAL: NCT02764073
Title: Bioimpedance Spectroscopy for the Evaluation of Heart Failure - a Comparison With Clinical Assessment, Lung Ultrasonography, Cardiac Biomarkers and Echocardiography
Brief Title: Bioimpedance Spectroscopy for the Evaluation of Heart Failure
Acronym: BIS-HF
Status: Completed | Type: Observational
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Professor Adrian Covic, Professor, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: BIS-HF
Record Dates: First submitted 2016-04-12; First posted 2016-05-06 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
Keywords: Heart failure; Bioimpedance; Lung ultrasonography
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bioimpedance spectroscopy — The technique involves attaching electrodes to the patient's forearm and ipsilateral ankle, with the patient in a supine position. The BCM® measures the body resistance and reactance to electrical currents of 50 discrete frequencies, ranging between 5 and 1000 kHz. Based on a fluid model using these resistances, the extracellular water (ECW), the intracellular water (ICW) and the total body water (TBW) are calculated. All calculations are automatically performed by the software of the BCM® device. Absolute fluid overload (AFO) is is defined as the difference between the expected patient's ECW under normal physiological conditions and the actual ECW, whereas the relative fluid overload (RFO) is defined as the absolute fluid overload AFO to ECW ratio.
  Other Names: BCM®Body Composition Monitor - Fresenius Medical Care D GmbH
Device: Lung Ultrasonography — Examinations will be performed in the supine position. Scanning of the anterior and lateral chest will be performed on both sides of the chest, from the second to the fourth (on the right side to the fifth) intercostal spaces, at parasternal to mid-axillary lines. B-lines will be recorded in each intercostal space and were defined as a hyperechoic, coherent US bundle at narrow basis going from the transducer to the limit of the screen. B-lines starting from the pleural line can be either localized or scattered to the whole lung and be present as isolated or multiple artifacts (with a distance 7 mm between 2 artifacts). The sum of B-lines produces a score reflecting the extent of lung water accumulation (0 being no detectable B-line).
Device: Echocardiography — All echocardiographic measurements will be carried out according to the recommendations of the American Society of Echocardiography by an observer unaware of the lung ultrasound and bioimpedance results. Echocardiographic evaluation will provide information about cardiac anatomy (e.g. volumes, geometry, mass) and function (e.g. left ventricular function and wall motion, valvular function, right ventricular function, pulmonary artery pressure, pericardium).

SUMMARY:
Despite impressive improvements in treatment strategies, heart failure (HF) morbidity and mortality remains substantially high worldwide. Pulmonary congestion is considered the leading cause for hospital admissions and death among patients with HF. Physical examination is crucial for titrating medical treatment in these patients, but despite a good specificity it is not sensitive enough to detect early elevated cardiac filling pressures.

The N-terminal pro-B-type natriuretic peptide (NT-proBNP) is a recognized powerful predictor for HF prognosis. Recently, cardiotrophin-1 and galectin-3 have been proposed as new relevant biomarkers for HF evaluation.

Echocardiography can be also used to noninvasively measure left ventricular filling pressures. Lung ultrasound (LUS) through interstitial B-line evaluation has been recently proposed as a bed-side, noninvasive tool to assess interstitial lung water. B-lines correlate with NT-proBNP and E/e' levels in patients with acute dyspnea, chronic HF or after a stress test. LUS can also identify clinically silent pulmonary edema, suggesting that it may complement clinical evaluation to improve hemodynamic profiling and treatment optimization.

Biompedance is a bedside method for total body fluid status assessment. It defines individual fluid status/compartments/overload on the basis of an individual's normal extracellular volume and body composition. Recent studies indicate that bioimpedance-derived fluid overload indices are independent predictors of mortality in renal failure patients.

To date, no study has evaluated bioimpedance performance for fluid assessment in HF patients. The investigators aim to cross-sectionally compare bioimpedance parameters with clinical evaluation, LUS, cardiac biomarkers, and echocardiographic characteristics, in a cohort of incident consecutive patients with HF. Two years patients' survival will be evaluated to propose the best evaluative algorithm and rank the various methods for prognostic significance.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years;
2. HF diagnosis regardless of cause as defined by the Framingham criteria and satisfying the European Society of Cardiology guidelines;

Exclusion Criteria:

1. metallic joint prostheses, cardiac stent or pacemakers, decompensated cirrhosis, pregnancy and limb amputations (due to bioimpedance technique limitations);
2. no prior diagnosis of pulmonary fibrosis (due to lung ultrasonography limitations);
3. absence of congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Heart Failure
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-05; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
The relationship between bioimpedance derived parameters (TBW, ICW, ECW, RFO), clinical assessment, lung congestion (as assessed by lung ultrasonography), echocardiography and different cardiac biomarkers. | 2 years

SECONDARY OUTCOMES:
The impact of baseline bioimpedance characteristics (TBW, ICW, ECW, RFO) on all-cause mortality. | 2 years
The impact of baseline bioimpedance characteristics (TBW, ICW, ECW, RFO) on fatal and non-fatal cardiovascular events. | 2 years
The impact of baseline bioimpedance characteristics (TBW, ICW, ECW, RFO) on hospitalizations. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. CI Parhon, Iași, Romania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Siriopol D, Popa R, Mihaila M, Rusu F, Sascau R, Statescu C, Catalina Z, Vasiliu V, Bucur A, Neamtu A, Siriopol I, Cianga P, Kanbay M, Covic A. Application of survival classification and regression tree analysis for identification of subgroups of risk in patients with heart failure and reduced left ventricular ejection fraction. Int J Cardiovasc Imaging. 2021 Jun;37(6):1853-1861. doi: 10.1007/s10554-021-02159-6. Epub 2021 Jan 16. PMID 33454896